CLINICAL TRIAL: NCT04781049
Title: Transperineal Laser Ablation Of Prostate Versus Transurethral Prostate Resection for Benign Prostatic Obstruction: A Randomized Clinical Trial
Brief Title: Transperineal Laser Ablation vs Transurethral Resection for Benign Prostatic Obstruction: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Carlo di Nancy Hospital (Other)
Collaborators: Elesta S.R.L. (Industry)
Responsible Party: Principal Investigator, Riccardo Bertolo, Assistant Professor, San Carlo di Nancy Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1580/CELazio1
Record Dates: First submitted 2021-02-22; First posted 2021-03-04 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Prostate Hyperplasia; Benign Prostatic Hyperplasia; Benign Prostatic Hypertrophy; Benign Prostatic Hypertrophy With Outflow Obstruction
Keywords: TPLA; TURP; BPH; BPO; LUTS
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPLA (Trans-Perineal Laser Ablation of Prostate) (Experimental): Participants who undergo Trans-Perineal Laser Ablation of Prostate
  Interventions: Procedure: Trans-Perineal Laser Ablation of Prostate
- TURP (Trans-Urethral Resection of Prostate) (Active Comparator): Participants who undergo the standard treatment, namely Trans-Urethral Resection of Prostate
  Interventions: Procedure: Trans-Urethral Resection of Prostate

INTERVENTIONS:
Procedure: Trans-Perineal Laser Ablation of Prostate — TPLA treatment will be performed using the EchoLaser EVO system (Elesta SpA - Calenzano, FI, Italy). EchoLaser EVO consists of four echolasers, a multi-source laser system with a wavelength of 1064nm and Echolaser Smart Interface (ESI), a treatment planning device for safely inserting introductor needles and optical fibers into prostate tissue. EchoLaser therapy is a micro-invasive percutaneous procedure that uses laser light transmitted through applicators (optical fibers) for a few minutes, causing a heating of the affected tissue to its irreversible damage in "situ", without the need to remove it. EchoLaser therapy, through flat-tip fibers, produces an ellipsoidal clotting area (area where the tissue has irreversible damage). EchoLaser therapy will be performed under ultrasound guidance.
  Arms: TPLA (Trans-Perineal Laser Ablation of Prostate)
Procedure: Trans-Urethral Resection of Prostate — TURP is the gold standard for the treatment of benign prostatic obstruction. It will be performed by using a bipolar energy resectoscope. The procedure will be carried out with patient in a lithotomic position.
  Arms: TURP (Trans-Urethral Resection of Prostate)

SUMMARY:
The primary objective of the study is to compare Trans-Perineal Laser Ablation of Prostate versus Trans-Urethral Resection of Prostate in the immediate impact on post-operative pain; in terms of relief in benign prostatic obstruction and preservation of the ejaculatory function in the short term (at 1, 3 and 6 months).

The secondary objective of the study is the evaluation of the long-term deobstructive effectiveness (12 months).

DETAILED DESCRIPTION:
Consecutive patients coming to our institution affected by benign prostatic obstruction (BPO) with indication to surgery and strong need of ejaculatory preservation will be enrolled in the present randomised controlled trial study after counseling. After an informed consent is obtained, uroflowmetry with calculation of the post-voiding residual volume (PVR), a transrectal ultrasonography to estimate prostate volume (PVol), the international prostate symptoms score (IPSS) questionnaire with quality of life (QoL) assessment, and the evaluation of the ejaculatory sexual function will be performed in all patients.

Trans-Perineal Laser Ablation of Prostate (TPLA) will be performed using the EchoLaser combined system (Elesta, Italy).

During the procedure, two 21G spinal needles are inserted transperineally in the peri-urethral area under ultrasound-guidance. By optical fibers, a maximum energy of 1800 J at a power of 3 Watts is delivered. If necessary, the fibers are eventually pulled-back. Immediately after the procedure, the patients will be asked to fill in the Visual Analogue Scale (VAS) for the assessment of the pain perceived. Perioperative data and postoperative data including assessment of ejaculatory function will be analyzed at different time points.

ELIGIBILITY:
Inclusion Criteria:

* signed written informed consent
* patient able to complete the Whole protocol
* IPSS score ≥ 10
* Maximum urinary flow rate < 15 ml/sec
* Prostate volume at preop. ultrasonography < 100 mL
* normal urinalysis (all of the above)

Exclusion Criteria:

* former prostate surgery
* prostate cancer (history)
* urethral stricture (history)
* Marion's disease (history)
* bladder stones
* median obstructive lobe, as defined by a > 1 cm of prostate abutting in the bladder lumen at ultrasonography
* neurological conditions potentially impacting on the bladder voiding (at least one of the above)

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study is investigating a novel micro-invasive treatment for benign prostatic obstruction. Thus, being male and having prostate in situ is mandatory.
Enrollment: 51 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2022-10-06 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analogue Scale (VAS) | Differences between preoperative and 4-hours postoperative
  Visual Analogue Scale. A standardized assessment of perceived pain. Scaled from a minimum of 0 to a maximum of 10 points.
Change in Ejaculatory function as assessed by the Male Sexual Health Questionnaire - Ejaculatory function domain (EJ-MSHQ) | Differences among preoperative status versus 1, 3, 6, 12 months after surgery
  EJ-MSHQ questionnaire will be used for a standardized assessment. Scaled from a minimum of 0 to a maximum of 25 points.
Changes in Sexual function as assessed by the International Index of Erectile Function Questionnaire (IIEF) | Differences among preoperative status versus 1, 3, 6, 12 months after surgery
  IIEF questionnaire will be used for a standardized assessment. Scaled from a minimum of 0 to a maximum of 25 points.

SECONDARY OUTCOMES:
Changes in International Prostate Symptom Score (IPSS) | Differences among preoperative status versus 1, 3, 6, 12 months after surgery
  Standardized Evaluation of the relief in prostate symptoms score. Scaled from a minimum of 0 to a maximum of 35 points.
Changes in Quality of Life (QoL) | Differences among preoperative status versus 1, 3, 6, 12 months after surgery
  Standardized Evaluation of the improvement in Quality of Life. Scaled from a minimum of 0 to a maximum of 6 points.
Changes in the maximum urinary flow rate at Uroflowmetry (Qmax) | Differences among preoperative status versus 1, 3, 6, 12 months after surgery
  objective improvement of maximum urinary flow rate at uroflowmetry. Measured in ml/s, scaled from 0 to the maximum of the distribution (usually no more than 50 ml/s)

CONTACTS AND LOCATIONS:
Overall Officials: Pierluigi Bove, MD, Principal Investigator — San Carlo di Nancy Hospital
Locations (1):
- San Carlo di Nancy Hospital, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No
The study will be subject of publication. The data will be available upon request.

REFERENCES:
- [Result] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, Van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-Committee of the International Continence Society. The standardisation of terminology in lower urinary tract function: report from the standardisation sub-committee of the International Continence Society. Urology. 2003 Jan;61(1):37-49. doi: 10.1016/s0090-4295(02)02243-4. No abstract available. PMID 12559262
- [Result] Martin SA, Haren MT, Marshall VR, Lange K, Wittert GA; Members of the Florey Adelaide Male Ageing Study. Prevalence and factors associated with uncomplicated storage and voiding lower urinary tract symptoms in community-dwelling Australian men. World J Urol. 2011 Apr;29(2):179-84. doi: 10.1007/s00345-010-0605-8. Epub 2010 Oct 21. PMID 20963421
- [Result] Gacci M, Corona G, Vignozzi L, Salvi M, Serni S, De Nunzio C, Tubaro A, Oelke M, Carini M, Maggi M. Metabolic syndrome and benign prostatic enlargement: a systematic review and meta-analysis. BJU Int. 2015 Jan;115(1):24-31. doi: 10.1111/bju.12728. Epub 2014 Aug 16. PMID 24602293
- [Result] Kupelian V, Wei JT, O'Leary MP, Kusek JW, Litman HJ, Link CL, McKinlay JB; BACH Survery Investigators. Prevalence of lower urinary tract symptoms and effect on quality of life in a racially and ethnically diverse random sample: the Boston Area Community Health (BACH) Survey. Arch Intern Med. 2006 Nov 27;166(21):2381-7. doi: 10.1001/archinte.166.21.2381. PMID 17130393
- [Result] Parsons JK. Benign Prostatic Hyperplasia and Male Lower Urinary Tract Symptoms: Epidemiology and Risk Factors. Curr Bladder Dysfunct Rep. 2010 Dec;5(4):212-218. doi: 10.1007/s11884-010-0067-2. Epub 2010 Sep 7. PMID 21475707
- [Result] Barry MJ, Fowler FJ Jr, O'Leary MP, Bruskewitz RC, Holtgrewe HL, Mebust WK, Cockett AT. The American Urological Association symptom index for benign prostatic hyperplasia. The Measurement Committee of the American Urological Association. J Urol. 1992 Nov;148(5):1549-57; discussion 1564. doi: 10.1016/s0022-5347(17)36966-5. PMID 1279218
- [Result] Siroky MB, Olsson CA, Krane RJ. The flow rate nomogram: II. Clinical correlation. J Urol. 1980 Feb;123(2):208-10. doi: 10.1016/s0022-5347(17)55859-0. PMID 7354519
- [Result] Biester K, Skipka G, Jahn R, Buchberger B, Rohde V, Lange S. Systematic review of surgical treatments for benign prostatic hyperplasia and presentation of an approach to investigate therapeutic equivalence (non-inferiority). BJU Int. 2012 Mar;109(5):722-30. doi: 10.1111/j.1464-410X.2011.10512.x. Epub 2011 Aug 22. PMID 21883855
- [Result] Perera M, Roberts MJ, Doi SA, Bolton D. Prostatic urethral lift improves urinary symptoms and flow while preserving sexual function for men with benign prostatic hyperplasia: a systematic review and meta-analysis. Eur Urol. 2015 Apr;67(4):704-13. doi: 10.1016/j.eururo.2014.10.031. Epub 2014 Nov 15. PMID 25466940
- [Result] de Rienzo G, Lorusso A, Minafra P, Zingarelli M, Papapicco G, Lucarelli G, Battaglia M, Ditonno P. Transperineal interstitial laser ablation of the prostate, a novel option for minimally invasive treatment of benign prostatic obstruction. Eur Urol. 2021 Jul;80(1):95-103. doi: 10.1016/j.eururo.2020.08.018. Epub 2020 Aug 28. PMID 32868137
- [Derived] Bertolo R, Iacovelli V, Cipriani C, Carilli M, Vittori M, Antonucci M, Maiorino F, Signoretti M, Petta F, Travaglia S, Panei M, Bove P. Ejaculatory function following transperineal laser ablation vs TURP for benign prostatic obstruction: a randomized trial. BJU Int. 2023 Jul;132(1):100-108. doi: 10.1111/bju.16008. Epub 2023 Mar 30. PMID 36917033